CLINICAL TRIAL: NCT05071963
Title: Neurovascular Product Surveillance Registry (INSPIRE) Pipeline™ Flex Embolization Device With Shield Technology™ Post Approval Study (PAS)
Brief Title: INSPIRE Pipeline™ Shield Post Approval Study
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT16056 (Shield PAS)
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Treatment of Intracranial Aneurysms — Embolization of aneurysms using the Pipeline™ Flex Embolization Device with Shield Technology™

SUMMARY:
The purpose of the Pipeline™ Flex Embolization Device with Shield Technology™ Post Approval Study (PAS) ("Pipeline™ Shield PAS") is to collect on-label use data in patients undergoing treatment for intracranial aneurysms (IA) using the Pipeline™ Flex Embolization Device with Shield Technology™ ("Pipeline™ Shield Device") in a real-world post approval setting within the United States.

DETAILED DESCRIPTION:
The INSPIRE Pipeline™ Shield Post Approval Study is an observational, prospective, multi-center, single-arm registry to collect on-label use data in patients undergoing treatment for intracranial aneurysms using the Pipeline™ Flex Embolization Device with Shield Technology™ according to the intended use.

The primary objective of this study is to evaluate the on-label use of the Pipeline™ Shield Device in patients undergoing treatment for intracranial aneurysms per institutional routine clinical care in a real-world post approval study setting in the U.S.

This study is conducted under the Product Surveillance Registry (NCT01524276) and is a sub-study to the therapy specific Neurovascular Product Surveillance Registry (NCT02988128).

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legally authorized representative (LAR) provides authorization and/or consent per institution and geographical requirements.
2. Patient is intended to receive or be treated with an eligible Medtronic product.
3. Patient is consented within the enrollment window of the therapy received, as applicable.
4. Patient or patient's legally authorized representative (LAR) has provided written informed consent using the IRB and Medtronic approved Informed Consent Form and agrees to comply with the study requirements. HIPAA/data protection authorization has been provided and signed by the patient (or patient's LAR).
5. Patient has already been selected for endovascular treatment of the target aneurysm with the Pipeline™ Shield Device as the appropriate treatment per the Pipeline™ Shield Device Instructions For Use (IFU).

Exclusion Criteria:

1. Patient who is, or is expected to be, inaccessible for follow-up.
2. Participation is excluded by local law.
3. Patient is currently enrolled or plans to enroll in a concurrent drug/device study that may confound the PSR results (i.e. no required intervention that could affect interpretation of all-around product safety and/or effectiveness).
4. Female patient who is known to be pregnant or is breastfeeding or wishes to become pregnant during participation in the study.
5. Patient is contraindicated for the device or procedure per the Pipeline™ Shield Device IFU.
6. The Investigator determined that the health of the patient may be compromised by the patient's enrollment.
7. Patient is enrolled or planning to participate in a potentially confounding drug or device trial during the course of this study. Co-enrollment in concurrent trials is only allowed when documented pre-approval was obtained from Medtronic.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring treatment for intracranial aneurysms with the market approved Pipeline™ Flex Embolization Device with Shield Technology™ device are eligible for the registry
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of the composite outcome (Occlusion of the target aneurysm, Significant parent artery stenosis, Retreatment of the target aneurysm) at 1 year post-procedure. | 1 year
  Incidence at 1-year post-procedure of complete occlusion of the target aneurysm, significant parent artery stenosis ≤ 50%, and no retreatment of the target aneurysm.

CONTACTS AND LOCATIONS:
Overall Officials: Harsh Sancheti, Study Director — Medtronic
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Yale New Haven Hospital, New Haven, Connecticut
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Endeavor Health - Evanston Hospital, Evanston, Illinois
  - Norton Healthcare, Louisville, Kentucky
  - Washington University in Saint Louis, St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
  - Montefiore Medical Center, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma (OU) University Medical Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Baylor Scott & White Research Institute, Dallas, Texas
  - University of Utah Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be available